CLINICAL TRIAL: NCT04623736
Title: Assessment of Smoking Cessation in a Publicly Available Cessation Smartphone Application
Brief Title: Smartphone Application Smoking Cessation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Cancer Institute (NCI) (NIH); ICF International (Unknown)
Responsible Party: Principal Investigator, Kara Wiseman, MPH, PhD, Assistant Professor, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3643
Record Dates: First submitted 2020-10-30; First posted 2020-11-10 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Tobacco Use
Keywords: Tobacco use; Smoking cessation; Smartphone applications; mHealth
MeSH Terms: conditions — Tobacco Use; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- quitSTART (Experimental)
  Interventions: Behavioral: quitSTART

INTERVENTIONS:
Behavioral: quitSTART — All participants will have access to the Smokefree.gov Initiative smoking cessation smartphone application, quitSTART. This app is available, at no cost, to anyone who owns a smartphone and is interested in quitting smoking. All smokers who download quitSTART are asked to provide basic information about themselves (e.g., age, sex, reason to quit smoking, triggers to smoke, when users typically smoke, how users plan to celebrate success, smoking frequency, age when started smoking regularly, ethnicity, race, cigarettes smoked per day), and set a quit date. Information about cessation and challenges to help support quitting are available, as well as games and tracking features. While using the app, users can proactively report cigarette cravings, if they slipped, if they are feeling "down" or feeling "great". If a user reports a craving, they have the option to mark the timing or location of the craving and request a reminder to resist future cravings at the same time or location.

SUMMARY:
The purpose of the study is to determine if using the smartphone application quitSTART can help people quit smoking and to understand how use of specific smartphone application features when trying to quit smoking is associated with success.

DETAILED DESCRIPTION:
Cigarette smoking is the leading cause of preventable death in the U.S. and causes multiple cancers. Approximately 34 million U.S. adults currently smoke cigarettes, but over half of all smokers attempt to quit smoking each year. However, only about 6% quit successfully, in part, because many smokers make unassisted quit attempts, due to the lack of accessibility of cessation programs. Mobile health (mHealth) smoking cessation programs delivered through smartphone applications ('apps') can potentially reach a large number of smokers in the U.S., as 81% of U.S. adult smokers own a smartphone. The National Cancer Institute hosts Smokefree.gov, a suite of free, publicly available smoking cessation resources. In addition to web based and text-messaging resources, Smokefree.gov launched the quitSTART smartphone app in 2013, which is a publicly available smoking cessation app.

Participants in this study will be asked to complete a pre-cessation assessment, then download, install, and try to quit smoking using the smoking cessation smartphone application, quitSTART. Participants will be asked to use quitSTART for 4 weeks. Participants will also be asked to complete online surveys 2 and 4 weeks after the start of the study. To understand how people are using quitSTART, the investigators will collect quitSTART usage data from all participants (for example, how often someone opens quitSTART during the study period and what specific features someone uses).

ELIGIBILITY:
Inclusion Criteria:

* Cigarette smoker
* Smoked at least 100 cigarettes
* Able to read and speak English
* Owns a smartphone
* 18 years of age or older
* USA resident

Exclusion Criteria:

* Not a cigarette smoker
* has not smoked at least 100 cigarettes
* Not able to read and speak English
* Does not own a smartphone
* Under 18 years of age
* Not a US resident
* Currently pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2021-05-12 (Actual); Study Completion 2021-06-10 (Actual)

PRIMARY OUTCOMES:
Self-reported 7-day smoking abstinence - 2 weeks | 2 weeks
  "Have you smoked a cigarette (even a puff) in the past 7 days?" self-reported by the participant
Self-reported 7-day smoking abstinence - 4 weeks | 4 weeks
  "Have you smoked a cigarette (even a puff) in the past 7 days?" self-reported by the participant

SECONDARY OUTCOMES:
Self-reported continuous smoking abstinence - 2 weeks | 2 weeks
  "In the last two weeks, have you smoked at all?" self-reported by the participant
Self-reported continuous smoking abstinence - 4 weeks | 4 weeks
  "In the last four weeks, have you smoked at all?" self-reported by the participant

CONTACTS AND LOCATIONS:
Overall Officials: Kara P Wiseman, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
If requested, a de-identified dataset will be available to other researchers after the study is completed.
Supporting Information: Study Protocol
Time Frame: After study completion

REFERENCES:
- [Derived] Siegel LN, Wiseman KP, Budenz A, Prutzman Y. Identifying Patterns of Smoking Cessation App Feature Use That Predict Successful Quitting: Secondary Analysis of Experimental Data Leveraging Machine Learning. JMIR AI. 2024 May 22;3:e51756. doi: 10.2196/51756. PMID 38875564